CLINICAL TRIAL: NCT00387751
Title: A Phase II, Pharmacokinetic (PK), Pharmacodynamic (PD) and Biological Correlative Study of the Efficacy and Safety of Dual Antiangiogenic Inhibition Using Bevacizumab and Sorafenib in Patients With Advanced Malignant Melanoma
Brief Title: Bevacizumab and Sorafenib in Treating Patients With Unresectable Stage III or Stage IV Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00134; NCI-2009-00134 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000502282; 05-25; 05-25 (Other: Cancer Therapy and Research Center at The UT Health Science Center at San Antonio); 7200 (Other: CTEP); P30CA054174 (NIH); U01CA069853 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Recurrent Melanoma; Stage III Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Sorafenib

ARMS (1):
- Arm I (Experimental): Patients receive oral sorafenib tosylate on days 1-5, 8-12, 15-19, and 22-26 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sorafenib Tosylate

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sorafenib Tosylate — Given orally
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with sorafenib works in treating patients with unresectable stage III or stage IV malignant melanoma. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and sorafenib may also stop the growth of melanoma by blocking blood flow to the tumor. Giving bevacizumab together with sorafenib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the clinical biologic activity of sorafenib tosylate and bevacizumab, defined as the sum of complete response, partial response, and prolonged stable disease for ≥ 16 weeks, in patients with unresectable stage III or stage IV malignant melanoma previously treated with at least 2 regimens of immunotherapy, cytokines, biologic therapy, or vaccine therapy or in previously untreated patients who are not appropriate candidates to receive aldesleukin-based treatment.

SECONDARY OBJECTIVES:

I. Evaluate the safety and tolerability of sorafenib tosylate and bevacizumab in these patients.

II. Evaluate the biologic activity of this regimen, in terms of time to progression, progression-free survival at 6 months, and overall survival, in these patients.

III. Describe significant pharmacokinetic interactions between bevacizumab and sorafenib tosylate.

IV. Characterize the pharmacodynamic relationships between the plasma concentration of sorafenib tosylate and bevacizumab and the effects of treatment on normal organ function and tumor tissue in these patients.

V. Identify predictive biomarkers of response to this regimen in these patients.

VI. Correlate changes in biological measurements with patient outcomes.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral sorafenib tosylate on days 1-5, 8-12, 15-19, and 22-26 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days in the absence of unacceptable toxicity or disease progression. Blood samples and tumor biopsies are obtained periodically for pharmacokinetic and pharmacodynamic studies. Samples are examined by liquid chromatography, mass spectrometry, immunohistochemistry, gene expression analysis, DNA mutation analysis, and genomic analysis for biological markers.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Criteria:

* No substance abuse
* Histologically or cytologically confirmed melanoma:

  * Unresectable (stage III) or metastatic (stage IV) disease
* Measurable disease, defined as >= 1 lesion that can be accurately and serially measured in >= 1 dimension as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan:

  * Cutaneous lesions measuring >= 1 cm will be considered measurable disease
* No primary ocular melanoma
* No active CNS metastatic brain or meningeal tumors:

  * Prior CNS disease allowed provided it was definitely treated >= 3 months ago AND there is no CNS disease by MRI or CT scan within the past 4 weeks
  * No residual disease
* Life expectancy > 12 weeks
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* WBC >= 3,000/mm3
* Absolute neutrophil count >= 1,500/mm3
* Platelet count >= 100,000/mm3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 2.5 times ULN
* Creatinine =< 1.5 times ULN OR creatinine clearance >= 60 mL/min
* Serum amylase < 1.5 times ULN OR lipase < 1.5 times ULN
* Urine protein:creatinine ratio < 1.0 OR urine protein < 1,000 mg by 24-hour urine collection
* No significant traumatic injury in the past 28 days
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for >= 6 months after completion of study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sorafenib tosylate and bevacizumab or other agents used in the study
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* None of the following medical conditions:

New York Heart Association class III-IV congestive heart failure; Cardiac arrhythmias, including atrial fibrillation if not adequately controlled; Active coronary artery disease or ischemia (e.g., unstable angina, cerebrovascular accident, transient ischemic attack, or myocardial infarction within the past 6 months); Uncontrolled hypertension

* None of the following medical conditions: Clinically significant peripheral vascular disease; Evidence of bleeding diathesis or coagulopathy
* No seizure disorder requiring medication (e.g., antiepileptics)
* No prior or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, or T1) or any cancer treated with intent to cure, rather than for palliation, < 3 years prior to study entry
* No more than 2 prior immunotherapy, cytokine therapy, biologic therapy, or vaccine therapy regimens (e.g., aldesleukin) for advanced or metastatic disease:
* (continued from above) Prior single-agent immunotherapy or combinations of immunotherapy as first treatment for advanced or metastatic disease allowed; Prior immunotherapy, cytokine therapy, biologic therapy, or vaccine therapy regimens in the adjuvant setting allowed
* No immunotherapy, cytokine therapy, biologic therapy, or vaccine therapy (e.g., aldesleukin) for advanced or metastatic disease within the past 4 weeks
* No prior organ allograft or stem cell transplantation
* No prior Ras-pathway inhibitors (including trastuzumab [Herceptin], farnesyl transferase inhibitors, or MEK inhibitors)
* No prior treatment with a drug that targets vascular endothelial growth factor (e.g., bevacizumab)
* No prior thalidomide or sorafenib tosylate
* No chemotherapy or radiotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C) and recovered:

Radiographic evidence of progression required for prior irradiated lesions

* No major surgical procedure or open biopsy within the past 28 days
* No Hypericum perforatum (St. John's wort) or rifampin within the past 3 weeks
* Concurrent full-dose anticoagulants (e.g., warfarin) with PT INR > 1.5 allowed provided the following criteria are met:

Patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin

* AND (continued from above) Patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent carbamazepine, phenytoin, or phenobarbital (drugs that induce CYP450 3A activity)
* No concurrent St. John's wort or rifampin
* No concurrent radiotherapy
* No concurrent major surgery
* No history of or suspected HIV infection or clinically significant hepatitis B or C
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No active clinically serious infections
* No dysphagia (difficulty swallowing)
* No medical, psychological, or social condition that may preclude study participation or evaluation of the study results

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muralidhar Beeram, Principal Investigator — Cancer Therapy and Research Center at The UT Health Science Center at San Antonio
Locations (1):
- Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Mahalingam D, Malik L, Beeram M, Rodon J, Sankhala K, Mita A, Benjamin D, Ketchum N, Michalek J, Tolcher A, Wright J, Sarantopoulos J. Phase II study evaluating the efficacy, safety, and pharmacodynamic correlative study of dual antiangiogenic inhibition using bevacizumab in combination with sorafenib in patients with advanced malignant melanoma. Cancer Chemother Pharmacol. 2014 Jul;74(1):77-84. doi: 10.1007/s00280-014-2479-8. Epub 2014 May 10. PMID 24817603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab and Sorafenib
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Sorafenib
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Clinical biologic activity of treatment, defined as the sum of complete response, partial response, and prolonged stable disease for ≥ 16 weeks, upon treatment with the combination of sorafenib and bevacizumab, in patients with advanced metastatic melanoma previously treated with immunotherapy or in previously untreated patients who are not appropriate candidates to receive IL-2-based treatment.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started of the appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 4 months
Measure: Number; unit: participants
Groups:
- Bevacizumab and Sorafenib: Bevacizumab was administered as a 5 mg/kg intravenous dose every 2 weeks. The dose was based on the patient's actual body weight; the dose recalculated if there was a weight change of >10% from baseline.
  Sorafenib was administered as a 200 mg oral dose twice daily, for 5 days every 7 days. Courses will be defined as 28-day treatment periods and will be repeated without interruption until development of progressive disease or development of serious drug related toxicities.
Arm/Group | Bevacizumab and Sorafenib
Number analyzed (Participants) | 14
participants | 11

2. Secondary Outcome: Safety and Tolerability
Description: Safety and tolerability of treatment, in terms of toxicity profile and incidence and rating of toxicity, according to NCI CTCAE v3.0 criteria.
Time Frame: 6 months
Population: Data were not collected
Groups:
- Safety and Tolerability: No data collected
Arm/Group | Safety and Tolerability
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival
Description: Determined by time to progression, progression-free suvival, and overall survival.
Time Frame: 6 months
Population: Data were not collected
Groups:
- Survival: No data collected
Arm/Group | Survival
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Bevacizumab and Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less